CLINICAL TRIAL: NCT01475812
Title: Daily Activities Are Sufficient to Induce Dynamic Pulmonary Hyperinflation and Dyspnea in Chronic Obstructive Pulmonary Disease Patients
Acronym: Hyperinflation
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Antonio A.M. Castro, Dr., Federal University of São Paulo
Other Study IDs: 0353/03
Record Dates: First submitted 2011-11-17; First posted 2011-11-21 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Dynamic Lung Hyperinflation; COPD Patients; Activities of Daily Livin.
Keywords: COPD; activities of daily living; pulmonary hyperinflation; exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Activities of Daily Living

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD hyperinflation
  Interventions: Other: Hyperinflation and ADL

INTERVENTIONS:
Other: Hyperinflation and ADL — Assessment of dynamic pulmonary hyperinflation during activities of daily living in COPD patients.

SUMMARY:
Introduction: Chronic obstructive pulmonary disease is a condition characterized by airflow limitation usually progressive and associated with inflammatory response of lung noxious particles. During a physical activity chronic obstructive pulmonary disease patients may develop dynamic pulmonary hyperinflation, increased dyspnea perception and decreased activity performance. The investigators hypothesize that some specific activities of daily living induce dynamic pulmonary hyperinflation in COPD patients. Objective: To measure dynamic lung hyperinflation and its influence in dyspnea perception in moderate and severe chronic obstructive pulmonary disease patients after activities of daily living. Methods: The investigators measured inspiratory capacity, dyspnea sensation, peripheral oxygen saturation, heart rate and respiratory rate in 19 chronic obstructive pulmonary disease (COPD) patients. These measurements were taken at rest and after daily living activities (such as going up and down a set of stairs, going up and down a ramp and sweeping and mopping a room).

ELIGIBILITY:
Inclusion Criteria:

* COPD patients diagnosed with moderate to very severe airway obstruction according to GOLD classification (9)
* clinical stability with no clinical exacerbation during the previous 30 days prior to the beginning of the study and to sign an informed consent form

Exclusion Criteria:

* Inability to perform the slow vital capacity maneuver
* excessive perceived dyspnea during the test
* arterial oxyhemoglobin saturation (SpO2) lower than 80% during activities and/or need of oxygen supplementation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators included 19 COPD patients (13 male) with moderate to very severe degree of airway obstruction, with a mean post bronchodilator forced expiratory volume in the first second (FEV1) of 48.7 ± 7.1% predicted and mean age of 64.1 ± 5.3.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2007-03

PRIMARY OUTCOMES:
Inspiratory capacity variability within the accomplishment of activities of daily living in COPD patients. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo/SP, Brazil